CLINICAL TRIAL: NCT02156167
Title: Clinical Validation of the Nucleus® CP810 Sound Processor for the Codacs™ System
Brief Title: Clinical Assessment of the External Sound Processor Worn by Patients Implanted With Codacs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL5441
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Severe to Profound Mixed Hearing Loss
Keywords: Otosclerosis, cochlear implant, acoustic stimulation
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP810 and Codacs™Test System (Experimental): Nucleus® CP810 Sound Processor for the Codacs™ system (CE marked) and Codacs™ Test System (CE marked)
  Interventions: Device: CP810 and Codacs™ system test

INTERVENTIONS:
Device: CP810 and Codacs™ system test — Nucleus® CP810 Sound Processor for the Codacs™ system (CE marked) and Codacs™ Test System (CE marked)

SUMMARY:
The purpose of this study is to evaluate the effect of the sound processor upgrade from the C-DACS investigational device Freedom sound processor to the Nucleus® CP810 sound processor for the Codacs™ system on the speech reception threshold in noise, to evaluate the usability of the Codacs™ Fitting Software, to evaluate the quality of life with the Nucleus® CP810 Sound Processor for the Codacs™ system, to collect long term data, to evaluate the acceptance criteria of the postoperative Codacs™ system test and to evaluate the usability of the Codacs™ Test System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects implanted with a Cochlear C-DACS investigational device

Exclusion Criteria:

* Participation in another medical device study
* Unwillingness or inability of the subject to comply with the study requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernst von Wallenberg, PhD, Study Director — Cochlear
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Lenarz T, Zwartenkot JW, Stieger C, Schwab B, Mylanus EA, Caversaccio M, Kompis M, Snik AF, D'hondt C, Mojallal H. Multicenter study with a direct acoustic cochlear implant. Otol Neurotol. 2013 Sep;34(7):1215-25. doi: 10.1097/MAO.0b013e318298aa76. PMID 23921930
- [Background] Lenarz T, Verhaert N, Desloovere C, Desmet J, D'hondt C, Gonzalez JC, Kludt E, Macias AR, Skarzynski H, Van de Heyning P, Vyncke C, Wasowski A. A comparative study on speech in noise understanding with a direct acoustic cochlear implant in subjects with severe to profound mixed hearing loss. Audiol Neurootol. 2014;19(3):164-74. doi: 10.1159/000358004. Epub 2014 Feb 18. PMID 24556905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Center contacted their patients, who received a Codacs device in another clinical trial by phone in October 2013
Groups:
- CP810: Nucleus® CP810 Sound Processor for the Codacs™ system (CE marked)
Period: Overall Study
Arm/Group | CP810
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CP810
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 66 [53 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Region of Enrollment [Number; unit: participants]
  Germany | 15

OUTCOME MEASURES:

1. Primary Outcome: Aided Speech Reception Threshold (SRT) in Noise Measured by Signal to Noise Ratio for 50% Correct Scores With the Oldenburger Sentence Test
Description: The Oldenburger Sentence test is an adaptive speech in noise test with a fixed noise level of typically 65 decibel (dB) sound pressure level (SPL) and a varying speech level, depending on how many words in a sentence were repeated correctly by the subject. The outcome of this test is the signal-to-noise ratio (SNR) at which 50% of words in the sentence list were correctly repeated by the subject. The SRT in noise with the Freedom sound processor at the initial study visit was compared to the SRT in noise with the CP810 at the 3 months follow-up at different measurement conditions.
  Speech and noise coming from the front (S0N0)- Speech coming from the front and noise coming from the implanted side (S0N90)- Everyday program (E): omnidirectional microphone- Noise program (N): directional microphone- Freedom Sound Processor (Freedom)- CP810 Sound Processor (CP810).
Time Frame: 3 months after initial upgraded fitting
Population: One subject did not visit the clinic for the 3 months follow-up, a second subject did not perform the speech in noise test at the 3 months follow-up due to tiredness
Measure: Mean (Standard Deviation); unit: dB SNR
Arm/Group | CP810
Number analyzed (Participants) | 13
dB SNR
  S0N0 - E - Freedom | -0.83 (2.04)
  S0N0 - E - CP810 | -1.45 (2.29)
  S0N90 - E - Freedom | 0.64 (2.92)
  S0N90 - E - CP810 | 0.89 (2.83)
  S0N0 - N - CP810 | -1.22 (1.69)
  S0N90 - N - CP810 | -3.78 (3.33)

ADVERSE EVENTS:
Time Frame: March 2014 to June 2015
Arm/Group | CP810
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less